CLINICAL TRIAL: NCT05397587
Title: An Open, Observational Study to Evaluate the Immunity Persistence of an Inactivated Enterovirus 71 Vaccine (Vero Cell) in Subjects Aged 6 to 71 Months
Brief Title: An Immunity Persistence Study of Enterovirus 71 Inactivated Vaccine (Vero Cell)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-EV71-3003-1
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group aged 6~23 months (Experimental): Up to 146 subjects aged 6~23 months and have received EV71 vaccine developed by Sinovac Biotech Co., Ltd will be collected blood samples at 36 months after full immunization and at the age of 72 months.
  Interventions: Biological: Experimental Vaccine
- Experimental Group aged 24~35 months (Experimental): Up to 128 subjects aged 24~35 months and have received EV71 vaccine developed by Sinovac Biotech Co., Ltd will be collected blood samples at 36 months after full immunization .
  Interventions: Biological: Experimental Vaccine
- Experimental Group aged 36~71 months (Experimental): 100 subjects aged 36~71 months and have received EV71 vaccine developed by Sinovac Biotech Co., Ltd will be collected blood samples at 36 months after full immunization .
  Interventions: Biological: Experimental Vaccine
- Control Group aged 36~71 months (Active Comparator): 100 subjects aged 36~71 months and have received EV71 vaccine developed by Institute of Medical Biology,Chinese Academy of Medical Sciences will be collected blood samples at 36 months after full immunization .
  Interventions: Biological: Control Vaccine

INTERVENTIONS:
Biological: Experimental Vaccine — The EV71 vaccine was manufactured by Sinovac Biotech Co., Ltd and inactivated EV71 virus antigen was no less than 3.0EU in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: Enterovirus Type 71 Vaccine（Vero Cell）, Inactivated
  Arms: Experimental Group aged 24~35 months; Experimental Group aged 36~71 months; Experimental Group aged 6~23 months
Biological: Control Vaccine — The EV71 vaccine was manufactured by Institute of Medical Biology,Chinese Academy of Medical Sciences ,and inactivated EV71 virus antigen was no less than 3.0EU in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: Enterovirus Type 71 Vaccine, Inactivated（Human Diploid Cell）
  Arms: Control Group aged 36~71 months

SUMMARY:
This is an open，observational and follow-up clinical trial based on the clinical trial of EV71 vaccine extended age group.The purpose of this study is to evaluate the immunity persistence of EV71 vaccine developed by Sinovac Biotech Co., Ltd in subjects aged 6 ~71 months after full immunization of two doses of vaccine.

DETAILED DESCRIPTION:
This study is an open,observational and follow-up clinical trial of EV71 vaccine based on the clinical trial of EV71 vaccine extended age group.The main purpose of this study is to evaluate the immunity persistence of EV71 vaccine developed by Sinovac Biotech Co., Ltd in subjects aged 6~71 months after full immunization of two doses of vaccine.In this study, a total of 474 subjects from the EV71 vaccine extended age clinical trial who received two doses of experimental or control vaccine and were enrolled in the PPS set，including 274 subjects aged 6~35 months (the maximum number of subjects aged 6-23 months is 146, and the maximum number of subjects aged 24-35 months is 128),100 subjects aged 36~71 months and were enrolled in experimental group(EV71 vaccine developed by Sinovac Biotech Co., Ltd) and 100 subjects aged 36~71 months and were enrolled in control group(EV71 vaccine developed by Institute of Medical Biology,Chinese Academy of Medical Sciences) will be enrolled .Blood samples will be collected from subjects aged 6-23 months at 36 months after full immunization and at the age of 72 months.Blood samples will be collected from subjects aged 24 to 35 months at 36 months after full immunization.Blood samples will be collected from subjects aged 36-71 months at 36 months after the full immunization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the EV71 vaccine extended age clinical trial who received two doses of experimental or control vaccine and were enrolled in the PPS set;
* Provide legal identification;
* Participants or guardians of the participants should be capable of understanding the written consent form and voluntarily participate in the clinical trial.

Exclusion Criteria:

* Vaccination history of vaccines containing EV71 antigen components other than the EV71 vaccine expanded age group clinical trial;
* History of hand, foot and mouth disease caused EV71;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 474 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The seroconversion rates (SCR) of EV71 neutralizing antibody of all enrolled subjects | At 36 months after full immunization
  The seroconversion rates (SCR) of EV71 neutralizing antibody of all subjects at 36 months after full immunization.
The seroconversion rates (SCR) of the EV71 neutralizing antibody of subjects aged 6-23 months | At the age of 72 months
  The seroconversion rates (SCR) of the EV71 neutralizing antibody of subjects aged 6-23 months at the age of 72months.
GMT of the EV71 neutralizing antibody of all enrolled subjects | At 36 months after full immunization
  GMT of the EV71 neutralizing antibody of all enrolled subjects at 36 months after full immunization.
GMT of the EV71 neutralizing antibody of subjects aged 6-23 months | At the age of 72 months
  GMT of the EV71 neutralizing antibody of subjects aged 6-23 months at the age of 72months.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Master, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention
Locations (1):
- Yun County Center for Disease Control and Prevention, Lincang, Yunnan, China